CLINICAL TRIAL: NCT01604343
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study of CNTO 136 (Sirukumab), a Human Anti-IL-6 Monoclonal Antibody, Administered Subcutaneously, in Subjects With Active Rheumatoid Arthritis Despite DMARD Therapy
Brief Title: A Study of CNTO 136 (Sirukumab), Administered Subcutaneously, in Patients With Active Rheumatoid Arthritis Despite Disease-Modifying Antirheumatic Drug (DMARD) Therapy (SIRROUND-D)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100866; CNTO136ARA3002 (Other: Janssen Research & Development, LLC); 2010-022242-24 (EudraCT Number); U1111-1135-6325 (Other: Universal Trial Number)
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Results first posted 2018-01-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Arthritis, Rheumatoid
Keywords: Active rheumatoid arthritis despite disease-modifying antirheumatic drug therapy; Sirukumab; Human Anti-IL-6 monoclonal antibody
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sirukumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- Placebo then Sirukumab 50 mg or Sirukumab 100 mg (Experimental)
  Interventions: Drug: Placebo; Drug: Sirukumab
- Sirukumab 100 mg (Experimental)
  Interventions: Drug: Sirukumab
- Sirukumab 50 mg + Placebo (Experimental)
  Interventions: Drug: Placebo; Drug: Sirukumab

INTERVENTIONS:
Drug: Placebo — Form=solution for injection, route=subcutaneous use; every 2 weeks from Week 0 through Week 50.
  Arms: Placebo then Sirukumab 50 mg or Sirukumab 100 mg
Drug: Placebo — Form=solution for injection, route=subcutaneous use; Weeks 2, 6, and every 4 weeks through Week 104.
  Arms: Sirukumab 50 mg + Placebo
Drug: Sirukumab — Type=exact, unit=mg, number=50 or 100, form=solution for injection, route=subcutaneous use; every 2 weeks for 100 mg and every 4 weeks for 50 mg, Week 52 through Week 104.
  Arms: Placebo then Sirukumab 50 mg or Sirukumab 100 mg
Drug: Sirukumab — Type=exact, unit=mg, number=100, form=solution for injection, route=subcutaneous use; Weeks 0, 2, and every 2 weeks through Week 104.
  Arms: Sirukumab 100 mg
Drug: Sirukumab — Type=exact, unit=mg, number=50, form=solution for injection, route=subcutaneous use; Weeks 0, 4, and every 4 weeks through Week 104.
  Arms: Sirukumab 50 mg + Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of sirukumab as measured by the reduction of the signs and symptoms of rheumatoid arthritis (RA) and inhibition of radiographic progression in patients with active RA who are unresponsive to treatment with disease-modifying antirheumatic drugs (DMARD).

DETAILED DESCRIPTION:
Patients will be randomly assigned to treatment groups, and they and study personnel will not know the identity of the treatments given. Some patients will receive a placebo, which resembles a medication, but does not contain an active substance. This helps to determine if the study agent is effective. Patients will receive placebo or sirukumab by injection under the skin. The expected duration of the study is 120 weeks, which includes 104 weeks of treatment. Participants who complete participation in the study will be eligible for inclusion into the long-term safety and efficacy study, if enrollment at a participating site is available to them. If they do not participate in the long-term study, they will continue into the safety follow-up for approximately 16 weeks. The placebo-controlled portion of the study is through Week 52, when placebo patients will cross over to one of two sirukumab dose regimens. Patient safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of rheumatoid arthritis (RA) for at least 3 months before screening
* Have moderately to severely active RA with at least 6 of 68 tender joints and 6 of 66 swollen joints, at screening and at baseline
* Have been unresponsive to single-agent or combination disease-modifying antirheumatic drugs (DMARD) therapy that includes methotrexate (MTX) or sulfasalazine (SSZ) due to lack of benefit after at least 12 weeks of DMARD, as assessed by the treating physician
* If using oral corticosteroids, must be on a stable dose equivalent to less than or equal to 10 mg/day of prednisone for at least 2 weeks prior to the first administration of study agent. If currently not using corticosteroids, must not have received oral corticosteroids for at least 2 weeks prior to the first administration of study agent
* If using non nonsteroidal anti-inflammatory drug (NSAIDs) or other analgesics for RA, must be on a stable dose for at least 2 weeks prior to the first administration of study agent
* If using non-biologic DMARD such as MTX, SSZ, hydroxychloroquine, chloroquine, or bucillamine, must be on a stable dose for at least 4 weeks prior to the first administration of study agent and should have no serious toxic side effects attributable to the DMARD

Exclusion Criteria:

* Has a history of intolerance to at least 2 or inadequate response to at least 1 anti-tumor necrosis factor alpha agent after 3 months of therapy
* Has received infliximab, golimumab, adalimumab, or certolizumab pegol within 3 months of the first study agent administration
* Has received etanercept or yisaipu within 6 weeks of the first study agent administration
* Has a history of intolerance to tocilizumab that precluded further treatment with it, or inadequate response to 3 months of tocilizumab (anti-IL-6 receptor) therapy
* Has used B-cell-depleting therapy (eg, rituximab) within 7 months of first study agent administration or have evidence during screening of abnormally low B cell level caused by previous B-cell depletion therapy
* Has used anakinra within 4 weeks of first study agent administration
* Has used any other biologic therapy for the treatment of RA within 3 months of the first study agent administration
* Has received intra-articular (IA), intramuscular (IM), or intravenous (IV) corticosteroids for RA, including adrenocorticotrophic hormone during the 4 weeks prior to first study agent administration-
* Has received leflunomide within 24 months before the first study agent administration and have not undergone a drug elimination procedure, unless the M1 metabolite is measured and is undetectable. If a drug elimination procedure is performed during screening, the M1 metabolite should be measured and found to be undetectable
* Has a history of cyclophosphamide or cytotoxic agent use
* Has received cyclosporine A, azathioprine, tacrolimus, mycophenolate mofetil, oral or parenteral gold, or D-penicillamine within 4 weeks of the first study agent administration
* Has received an investigational drug (including investigational vaccines) or used an investigational medical device within 3 months or 5 half lives, whichever is longer, before the first study agent administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1670 (Actual)
Dates: Start 2012-08-15 (Actual); Primary Completion 2015-09-02 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (156):
- United States (48):
  - Glendale, Arizona
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Covina, California
  - El Cajon, California
  - Glendale, California
  - Hemet, California
  - Huntington Beach, California
  - La Jolla, California
  - La Palma, California
  - Whittier, California
  - Aventura, Florida
  - Brandon, Florida
  - Daytona Beach, Florida
  - Lake Mary, Florida
  - Naples, Florida
  - Palm Harbor, Florida
  - Tampa, Florida
  - Zephyrhills, Florida
  - Indianapolis, Indiana
  - Cedar Rapids, Iowa
  - Bowling Green, Kentucky
  - Monroe, Louisiana
  - Wheaton, Maryland
  - Eagan, Minnesota
  - Springfield, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Plainview, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Middleburg Heights, Ohio
  - Edmond, Oklahoma
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Wyomissing, Pennsylvania
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Mesquite, Texas
  - Kennewick, Washington
  - Beckley, West Virginia
  - Clarksburg, West Virginia
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Canada (5):
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Ottawa, Ontario
  - Burlington
  - Edmonton
- Chile (3):
  - Rancagua
  - Santiago
  - Valdivia
- Colombia (3):
  - Bogotá
  - Chía
  - Medellín
- Croatia (3):
  - Osijek
  - Rijeka
  - Zagreb
- Japan (30):
  - Ayauta-Gun
  - Bunkyō City
  - Fukuoka
  - Higashihiroshima
  - Izumo
  - Kagoshima
  - Katō
  - Kawagoe
  - Kita-Gun
  - Kumamoto
  - Kurume
  - Miyazaki
  - Nagano
  - Nagasaki
  - Nagoya
  - Osaka
  - Sapporo
  - Sasebo
  - Shimonoseki
  - Shimotsuke
  - Shinjuku-Ku
  - Sumida-Ku
  - Takaoka,Toyama
  - Takasaki
  - Tokorozawa
  - Tokushima
  - Tomishiro
  - Tsu
  - Ureshino
  - Yokohama
- Lithuania (4):
  - Alytus
  - Kaunas
  - Klaipėda
  - Šiauliai
- Malaysia (2):
  - Kuala Lumpur
  - Kuching
- Mexico (9):
  - Cuernavaca
  - Guadalajara
  - Juárez
  - Mexicali
  - Mexico City
  - Mérida
  - México
  - Morelia
  - San Luis de Potosi
- Poland (7):
  - Bialystok
  - Bydgoszcz
  - Elblag
  - Lublin
  - Poznan
  - Ustroń
  - Warsaw
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Iași
- Russia (10):
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Orenburg
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Ulyanovsk
  - Yaroslavl
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Niška Banja
- South Africa (3):
  - Cape Town
  - Port Elizabeth
  - Pretoria
- South Korea (10):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Incheon
  - Jeonju
  - Namdong-Gu
  - Seongnam-si
  - Seoul
  - Suwon
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- Ukraine (8):
  - Donetsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Odesa
  - Sympheropol
  - Vinnytsia
  - Zaporizhzhia

REFERENCES:
- [Derived] Takeuchi T, Thorne C, Karpouzas G, Sheng S, Xu W, Rao R, Fei K, Hsu B, Tak PP. Sirukumab for rheumatoid arthritis: the phase III SIRROUND-D study. Ann Rheum Dis. 2017 Dec;76(12):2001-2008. doi: 10.1136/annrheumdis-2017-211328. Epub 2017 Aug 30. PMID 28855173

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2746 participants were screened of which 1670 participants were randomized and received at least one administration of study treatment.
Groups:
- Placebo: Participants received Placebo subcutaneously (SC) every 2 weeks (q2w) from Week (W) 0 up to Week 50. Participants who met early escape (EE) criteria at Week 18, or late escape (LE) at Week 40, or cross-over (CO) at Week 52 were rerandomized to receive sirukumab 50 or 100 mg through Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
- Placebo to 50 mg q4w Due to EE/LE/CO: Participants who were assigned to placebo group and who met EE at Week 18 or LE at Week 40 or CO at Week 52 were re-randomized to receive subcutaneous (SC) sirukumab 50 mg dose regimen q4w up to Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
- Sirukumab 50 mg q4w: All participants received 50 mg of sirukumab subcutaneously every 4 weeks (q4w) for 104 weeks and in between placebo SC injections was received at Weeks 2, 6, and q4w through week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
- Placebo to 100 mg q2w Due to EE/LE/CO: Participants who were assigned to placebo group and who met EE at Week 18 or LE at Week 40 or CO at Week 52 were re-randomized to receive subcutaneous (SC) sirukumab 100 mg dose regimen q2w up to Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
- Sirukumab 100 mg q2w: All participants received 100 mg of sirukumab SC injections at Weeks 0, 2, and q2w through Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
Period: Prior to W52 Administration(Through W52)
Arm/Group | Placebo | Placebo to 50 mg q4w Due to EE/LE/CO | Sirukumab 50 mg q4w | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 100 mg q2w
Started | 556 | 0 | 557 | 0 | 557
Participants Re-randomized at Week 18 | 187 (Out of 187, 95 were re-randomized to sirukumab 50 mg and 92 were re-randomized to 100 mg group.) | 0 | 0 | 0 | 0
Participants Re-randomized at Week 40 | 24 (Out of 24, 12 were re-randomized to sirukumab 50 mg and 12 were re-randomized to 100 mg group.) | 0 | 0 | 0 | 0
Completed | 458 | 0 | 481 | 0 | 470
Not Completed | 98 | 0 | 76 | 0 | 87
Not completed — Lost to Follow-up | 5 | 0 | 4 | 0 | 3
Not completed — Withdrawal by Subject | 19 | 0 | 12 | 0 | 16
Not completed — Adverse Event | 25 | 0 | 41 | 0 | 42
Not completed — Death | 5 | 0 | 2 | 0 | 4
Not completed — Lack of Efficacy | 24 | 0 | 5 | 0 | 14
Not completed — Physician Decision | 4 | 0 | 1 | 0 | 2
Not completed — Pregnancy | 1 | 0 | 1 | 0 | 0
Not completed — Other | 15 | 0 | 10 | 0 | 6
Period: Week 52 to Week 104
Arm/Group | Placebo | Placebo to 50 mg q4w Due to EE/LE/CO | Sirukumab 50 mg q4w | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 100 mg q2w
Started | 0 | 243 (Participants re-randomized at Week 18 (95), 40 (12) and 52 were included) | 481 | 241 (Participants re-randomized at Week 18 (92), 40 (12) and 52 were included) | 470
Treated | 0 | 242 | 481 | 241 | 470
Completed | 0 | 200 | 414 | 195 | 429
Not Completed | 0 | 43 | 67 | 46 | 41
Not completed — Lost to Follow-up | 0 | 2 | 4 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 7 | 12 | 8 | 4
Not completed — Adverse Event | 0 | 12 | 26 | 21 | 27
Not completed — Death | 0 | 4 | 2 | 5 | 0
Not completed — Lack of Efficacy | 0 | 6 | 11 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 1 | 2 | 1
Not completed — Other | 0 | 11 | 11 | 6 | 3
Period: Safety Follow-up Period (Week 104-120)
Arm/Group | Placebo | Placebo to 50 mg q4w Due to EE/LE/CO | Sirukumab 50 mg q4w | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 100 mg q2w
Started | 109 | 27 | 105 | 36 | 114
Safety Population | 109 | 26 | 105 | 36 | 114
Completed | 79 | 20 | 72 | 26 | 85
Not Completed | 30 | 7 | 33 | 10 | 29
Not completed — Lost to Follow-up | 3 | 1 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 12 | 4 | 11 | 3 | 14
Not completed — Other | 15 | 2 | 20 | 6 | 14

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received Placebo subcutaneously (SC) every 2 weeks (q2w) from Week 0 up to Week 50. Participants who met early escape (EE) criteria at Week 18, or late escape (LE) at Week 40, or cross-over (CO) at Week 52 were rerandomized to receive sirukumab 50 or 100 mg through Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
- Total: Total of all reporting groups
Arm/Group | Placebo | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w | Total
Number analyzed (Participants) | 556 | 557 | 557 | 1670
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (11.85) | 52.9 (11.8) | 53 (11.31) | 52.9 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 436 | 447 | 452 | 1335
  Male | 120 | 110 | 105 | 335
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 5 | 7 | 6 | 18
  Canada | 4 | 4 | 3 | 11
  Chile | 23 | 21 | 24 | 68
  Colombia | 17 | 13 | 11 | 41
  Croatia | 4 | 4 | 2 | 10
  Japan | 56 | 58 | 54 | 168
  Lithuania | 32 | 31 | 35 | 98
  Malaysia | 5 | 1 | 1 | 7
  Mexico | 33 | 41 | 41 | 115
  Poland | 64 | 51 | 54 | 169
  Republic of Korea | 21 | 16 | 31 | 68
  Romania | 3 | 6 | 6 | 15
  Russian Federation | 61 | 67 | 73 | 201
  Serbia | 52 | 47 | 45 | 144
  South Africa | 40 | 34 | 26 | 100
  Taiwan, Province of China | 5 | 14 | 5 | 24
  Ukraine | 50 | 50 | 52 | 152
  United States | 81 | 92 | 88 | 261

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response at Week 16
Description: ACR 20 response is greater than or equal to (>=) 20 percent (%) improvement in both tender joint count (68) and swollen joint count (66) and >= 20% improvement in 3 of following 5 assessments:Participant's assessment of pain using visual analog scale (VAS) (0-10 scale, 0=no pain and 10=worst possible pain),Participant's global assessment of disease activity by using VAS (scale ranges from 0 to 10, [0 = very well to 10 = very poor]), Physician's global assessment of disease activity using VAS (scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), Participant's assessment of physical function as measured by Health Assessment Questionnaire-Disability Index (HAQ-DI) (scale ranges from 0= no difficulty to 3= inability to perform a task in that area), and Serum C-reactive protein (CRP). Participants were analyzed according to randomized treatment groups they were assigned, regardless of treatments they actually received. Here, TF= treatment failure.
Time Frame: Week 16
Population: Full analysis set included all randomized participants. Participants were set to non-responders if meeting TF criteria prior to week 16 or having data missing.
Measure: Number; unit: Percentage of Participants
Groups:
- Sirukumab 50 mg: Participants received 50 mg of sirukumab subcutaneously every 4 weeks (q4w) for 104 weeks and in between placebo SC injections was received at Weeks 2, 6, and q4w through Week 104.
- Sirukumab 100 mg: Participants received 100 mg of sirukumab SC injections at Weeks 0, 2, and q2w through Week 104.
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants | 26.4 | 54.8 | 53.5
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 28.4, 95% CI 2-sided [22.8 to 33.8]
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 27.1, 95% CI 2-sided [21.6 to 32.6]

2. Primary Outcome: Change From Baseline in Van Der Heijde-modified Sharpe (vdH-S) Score at Week 52
Description: The van der Heijde-modified Sharpe (vdH-S) score is defined as a measurement of progression in structural damage. It is the sum of joint erosion (32 joints of the hands and 12 joints of the feet) score and joint space narrowing (JSN) (30 joints of the hands and 12 joints of the feet) score. The joint erosion assessment is scored according to the surface area involved, from 0 to 5, with 0 indicating no erosion and 5 indicating complete collapse of bone whereas the JSN assessment including subluxation, is scored from 0 (normal) to 4 (bony ankylosis or complete luxation). The total score ranges from 0 (best) to 448 (worst) with higher scores indicating more joint damage. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received. Here, EE= early escape.
Time Frame: Baseline, Week 52
Population: Efficacy full analysis set (radiographic endpoints) had randomized participants received at least 1 (partial/complete) dose of study drug with non-missing baseline vdH-S score. It was based on imputed value by EE Rules: set scores after EE missing for placebo arm; and then missing data rules in all treatment arms using linear extrapolation method.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 550 | 553 | 551
Units on a Scale | 3.69 (9.245) | 0.50 (2.961) | 0.46 (3.258)
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p < 0.001, van der waerden ANOVA
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, van der waerden ANOVA

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) score is an evaluation of the functional status for a participant. The 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range: 0-3 where 0 = least difficulty and 3 = extreme difficulty. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 24
Population: Full analysis set included all randomized participants. Last Observation Carried Forward (LOCF) method was used to impute missing values. Last Observation at or prior EE was used to replace the data after EE for participants who met EE criteria.
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Units on Scale | -0.2179 (0.53081) | -0.4262 (0.57631) | -0.4610 (0.56784)
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Square (LS) mean difference = -0.2260, 95% CI 2-sided [-0.29 to -0.17]
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.2560, 95% CI 2-sided [-0.32 to -0.20]

4. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 50 Response at Week 24
Description: An American College of Rheumatology (ACR) 50 response is defined as >= 50 % improvement in both tender joint count (68 joints) and swollen joint count (66 joints) and >= 50% improvement in 3 of the following 5 assessments: Participant's assessment of pain using VAS (0-10 scale, 0=no pain and 10=worst possible pain), Participant's global assessment of disease activity by using VAS (the scale ranges from 0 to 10, [0 = very well to 10 = very poor]), Physician's global assessment of disease activity using VAS (the scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), Participant's assessment of physical function as measured by HAQ-DI (the scale ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area), and Serum CRP. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 24
Population: Full analysis set included all randomized participants. Participants were set to non-responders if meeting EE or TF criteria prior to week 24 or having data missing.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants | 12.4 | 30.2 | 33.2
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 17.8, 95% CI 2-sided [13.1 to 22.4]
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 20.8, 95% CI 2-sided [16.1 to 25.6]

5. Secondary Outcome: Percentage of Participants With Disease Activity Index Score 28 (DAS28) (C-reactive Protein (CRP) Remission at Week 24
Description: The DAS28 based on C-Reactive Protein (CRP) is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. The Disease Activity Index Score 28 (DAS28) C-reactive protein (CRP) remission is defined as a DAS28 (CRP) value of less than 2.6 at a visit. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 24
Population: Full analysis set included all randomized participants. Participants were set to not achieving DAS28 remission if meeting EE or TF criteria prior to week 24 or having data missing.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants | 5.6 | 26.0 | 25.5
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 20.5, 95% CI 2-sided [16.4 to 24.6]
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 19.9, 95% CI 2-sided [15.8 to 24.0]

6. Secondary Outcome: Percentage of Participants With Major Clinical Response (MCR) at Week 52
Description: MCR- participant achieving ACR 70 response for 6 continuous months (24 weeks) in the study period (i.e., through Week 52). An ACR 70 response is defined as >= 70% improvement in both tender joint count (68 joints) and swollen joint count (66 joints) and >= 70% improvement in 3 of the following 5 assessments Participant's assessment of pain using VAS (0-10 scale, 0=no pain and 10=worst possible pain), Participant's global assessment of disease activity by using VAS (scale ranges from 0 to 10, [0 = very well to 10 = very poor]), Physician's global assessment of disease activity using VAS (scale ranges from 0 to 10, [0=no arthritis to 10=extremely active arthritis]), Participant's assessment of physical function as measured by HAQ-DI (scale ranges from 0= no difficulty, to 3= inability to perform a task in that area) and Serum CRP. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 52
Population: Full analysis set was defined as all randomized participants. Participants were set to non-responders if meeting EE, LE or TF criteria prior to week 52 or having data missing.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants | 1.8 | 5.4 | 9.0
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 3.6, 95% CI 2-sided [1.4 to 5.8]
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 7.2, 95% CI 2-sided [4.6 to 9.8]

7. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response Through Week 52
Description: An ACR 20 response is defined as >= 20 % improvement in both tender joint count (68 joints) and swollen joint count (66 joints) and >= 20% improvement in 3 of the following 5 assessments: Participant's assessment of pain using VAS (0-10 scale, 0=no pain and 10=worst possible pain), Participant's global assessment of disease activity by using VAS (the scale ranges from 0 to 10, [0 = very well to 10 = very poor]), Physician's global assessment of disease activity using VAS (the scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), Participant's assessment of physical function as measured by HAQ-DI (the scale ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area), and Serum CRP. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 18, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Full analysis set included all randomized participants. Participants were set to non-responders after meeting EE, LE or TF criteria (whichever is earliest) or if having data missing.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 7.4 | 18.3 | 15.4
  Week 4 | 14.2 | 36.3 | 33.8
  Week 6 | 20.3 | 45.8 | 46.9
  Week 8 | 25.9 | 47.2 | 51.3
  Week 12 | 27.3 | 53.1 | 53.3
  Week 18 | 29.3 | 54.4 | 56.9
  Week 20 | 29.5 | 53.7 | 52.8
  Week 24 | 27.0 | 53.7 | 56.0
  Week 28 | 31.5 | 53.1 | 57.3
  Week 32 | 29.5 | 53.3 | 56.7
  Week 36 | 28.4 | 54.0 | 58.2
  Week 40 | 28.8 | 53.3 | 53.3
  Week 44 | 27.7 | 49.2 | 54.0
  Week 48 | 26.8 | 50.1 | 54.8
  Week 52 | 26.6 | 49.9 | 54.8

8. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 50 Response
Description: An ACR 50 response is defined as >= 50 % improvement in both tender joint count (68 joints) and swollen joint count (66 joints) and >= 50% improvement in 3 of the following 5 assessments: Participant's assessment of pain using VAS (0-10 scale, 0=no pain and 10=worst possible pain), Participant's global assessment of disease activity by using VAS (the scale ranges from 0 to 10, [0 = very well to 10 = very poor]), Physician's global assessment of disease activity using VAS (the scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), Participant's assessment of physical function as measured by HAQ-DI (the scale ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and Serum CRP. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 28, 32, 36, 40, 44, 48 and 52
Population: Full analysis set was defined as all randomized participants. Participants were set to non-responders after meeting EE, LE or TF criteria (whichever is earliest) or if having data missing.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 1.1 | 3.2 | 2.0
  Week 4 | 2.5 | 9.2 | 9.9
  Week 6 | 4.1 | 15.6 | 14.0
  Week 8 | 7.7 | 20.3 | 18.9
  Week 12 | 10.1 | 24.6 | 28.0
  Week 16 | 10.8 | 30.0 | 26.2
  Week 18 | 11.7 | 31.2 | 31.2
  Week 20 | 13.5 | 32.7 | 33.4
  Week 28 | 15.1 | 31.6 | 33.0
  Week 32 | 14.0 | 33.6 | 35.0
  Week 36 | 12.2 | 33.4 | 34.5
  Week 40 | 13.3 | 31.1 | 33.4
  Week 44 | 14.2 | 31.4 | 33.9
  Week 48 | 14.4 | 32.9 | 34.8
  Week 52 | 13.8 | 30.3 | 35.5

9. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 70 Response Through Week 52
Description: An ACR 70 response is defined as >= 70 % improvement in both tender joint count (68 joints) and swollen joint count (66 joints) and >= 70% improvement in 3 of the following 5 assessments: Participant's assessment of pain using VAS (0-10 scale, 0=no pain and 10=worst possible pain), Participant's global assessment of disease activity by using VAS (the scale ranges from 0 to 10, [0 = very well to 10 = very poor]), Physician's global assessment of disease activity using VAS (the scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), Participant's assessment of physical function as measured by HAQ-DI (the scale ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and Serum CRP. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 0.4 | 0.7 | 0.4
  Week 4 | 0.5 | 2.0 | 3.1
  Week 6 | 1.6 | 4.7 | 4.5
  Week 8 | 1.6 | 7.2 | 7.2
  Week 12 | 3.1 | 10.4 | 10.6
  Week 16 | 4.0 | 13.5 | 13.5
  Week 18 | 4.3 | 12.6 | 14.7
  Week 20 | 4.0 | 13.1 | 16.0
  Week 24 | 3.4 | 14.9 | 16.3
  Week 28 | 5.2 | 16.0 | 16.5
  Week 32 | 4.7 | 17.4 | 17.2
  Week 36 | 4.7 | 15.8 | 16.2
  Week 40 | 5.0 | 16.9 | 17.6
  Week 44 | 5.2 | 16.3 | 17.1
  Week 48 | 6.8 | 18.5 | 17.8
  Week 52 | 5.4 | 16.5 | 18.5

10. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 90 Response Through Week 52
Description: An ACR 90 response is defined as >= 90 percent (%) improvement in both tender joint count (68 joints) and swollen joint count (66 joints) and >= 90% improvement in 3 of the following 5 assessments: Participant's assessment of pain using VAS (0-10 scale, 0=no pain and 10=worst possible pain), Participant's global assessment of disease activity by using VAS (the scale ranges from 0 to 10, [0 = very well to 10 = very poor]), Physician's global assessment of disease activity using VAS (the scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), Participant's assessment of physical function as measured by HAQ-DI (the scale ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and Serum CRP. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 0 | 0 | 0
  Week 4 | 0 | 0.2 | 0.2
  Week 6 | 0.2 | 0.2 | 0.2
  Week 8 | 0.2 | 1.1 | 0.5
  Week 12 | 0.5 | 2.2 | 1.8
  Week 16 | 0.9 | 2.5 | 2.9
  Week 18 | 1.1 | 2.5 | 2.5
  Week 20 | 0.5 | 3.6 | 4.1
  Week 24 | 0.5 | 3.4 | 5.2
  Week 28 | 0.4 | 4.5 | 4.7
  Week 32 | 1.1 | 4.1 | 5.7
  Week 36 | 0.9 | 4.8 | 5.4
  Week 40 | 0.7 | 5.4 | 6.1
  Week 44 | 0.5 | 5.0 | 6.6
  Week 48 | 0.7 | 4.7 | 6.3
  Week 52 | 1.3 | 4.5 | 5.6

11. Secondary Outcome: Percentage of Participants With Disease Activity Index Score 28 (DAS28) C-reactive Protein (CRP) Response Through Week 52
Description: DAS28 based on C-Reactive Protein (CRP), a statistically derived index combining tender joints (28), swollen joints (28), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both upper right extremity and upper left extremity as well as knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. Good responders: improvement from baseline greater than (>) 1.2 with DAS28 less than or equal to (<=) 3.2; moderate responders: improvement from baseline >1.2 with DAS28 >3.2 to <=5.1 or improvement from baseline >0.6 to <=1.2 with DAS28 <=5.1; non-responders: improvement from baseline <=0.6 or improvement from baseline >0.6 and <=1.2 with DAS28 >5.1. Participants were analyzed according to randomized treatment groups they were assigned to, regardless of treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 18.5 | 72.0 | 72.4
  Week 4 | 28.1 | 80.1 | 78.3
  Week 6 | 36.7 | 82.4 | 80.3
  Week 8 | 38.5 | 81.7 | 81.3
  Week 12 | 43.7 | 83.3 | 81.3
  Week 16 | 42.6 | 80.4 | 79.5
  Week 18 | 41.5 | 79.7 | 79.4
  Week 20 | 41.5 | 73.8 | 72.5
  Week 24 | 37.9 | 71.5 | 72.2
  Week 28 | 41.2 | 69.7 | 72.2
  Week 32 | 41.4 | 68.2 | 70.6
  Week 36 | 39.7 | 67.7 | 69.8
  Week 40 | 39.2 | 66.8 | 67.9
  Week 44 | 37.6 | 63.2 | 64.6
  Week 48 | 36.7 | 61.9 | 64.6
  Week 52 | 35.6 | 62.5 | 64.3

12. Secondary Outcome: Change From Baseline in Disease Activity Index Score 28 (DAS28) C-reactive Protein (CRP) Through Week 52
Description: The DAS28 based on C-Reactive Protein (CRP) is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. A negative change from baseline in DAS28 (CRP) (that is, a decrease from baseline) indicates improvement from baseline. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: Full analysis set included all randomized participants. Last Observation Carried Forward (LOCF) method was used to impute missing values. Last Observation at or prior EE/LE was used to replace the data after EE/LE for participants who met EE/LE criteria.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Units on a Scale
  Change at Week 2 | -0.319 (0.7677) | -1.316 (0.7776) | -1.284 (0.7605)
  Change at Week 4 | -0.515 (0.9287) | -1.638 (0.9759) | -1.627 (0.9529)
  Change at Week 6 | -0.707 (1.0599) | -1.886 (1.0622) | -1.888 (1.0340)
  Change at Week 8 | -0.754 (1.1013) | -2.016 (1.1183) | -2.031 (1.1138)
  Change at Week 12 | -0.881 (1.1727) | -2.187 (1.1995) | -2.185 (1.1950)
  Change at Week 16 | -0.908 (1.2834) | -2.264 (1.2443) | -2.282 (1.2283)
  Change at Week 18 | -0.895 (1.2986) | -2.286 (1.2690) | -2.335 (1.2314)
  Change at Week 20 | -0.920 (1.2973) | -2.367 (1.3368) | -2.380 (1.3158)
  Change at Week 24 | -0.912 (1.3180) | -2.356 (1.3599) | -2.402 (1.3048)
  Change at Week 28 | -0.979 (1.3752) | -2.417 (1.4068) | -2.440 (1.3245)
  Change at Week 32 | -1.010 (1.3904) | -2.451 (1.4141) | -2.479 (1.3304)
  Change at Week 36 | -1.019 (1.4020) | -2.461 (1.3951) | -2.497 (1.3231)
  Change at Week 40 | -0.985 (1.4054) | -2.462 (1.4180) | -2.459 (1.3901)
  Change at Week 44 | -0.994 (1.4117) | -2.442 (1.4364) | -2.477 (1.4381)
  Change at Week 48 | -1.026 (1.4755) | -2.482 (1.4630) | -2.488 (1.3783)
  Change at Week 52 | -0.992 (1.4431) | -2.491 (1.4305) | -2.476 (1.4109)

13. Secondary Outcome: Percentage of Participants With Disease Activity Index Score 28 (DAS28) (C-reactive Protein (CRP) Remission Through Week 52
Description: as for outcome 5
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 28, 32, 36, 40, 44, 48 and 52
Population: Full analysis set included all randomized participants. Participants were set to not achieving DAS28 remission after meeting EE, LE or TF criteria (whichever is earliest) or if having data missing.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 0.5 | 2.5 | 2.7
  Week 4 | 1.6 | 7.9 | 9.3
  Week 6 | 3.1 | 10.2 | 12.6
  Week 8 | 3.2 | 13.6 | 17.8
  Week 12 | 4.3 | 18.3 | 19.6
  Week 16 | 5.8 | 21.2 | 21.9
  Week 18 | 6.1 | 22.8 | 23.7
  Week 20 | 5.8 | 26.4 | 25.5
  Week 28 | 7.7 | 27.5 | 27.1
  Week 32 | 7.7 | 29.6 | 28.4
  Week 36 | 8.5 | 29.1 | 28.0
  Week 40 | 7.2 | 27.8 | 27.3
  Week 44 | 8.5 | 28.2 | 27.5
  Week 48 | 9.0 | 29.6 | 30.2
  Week 52 | 8.8 | 30.0 | 29.1

14. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Score Through Week 52
Description: The SDAI score is a derived score combining tender joints (28 joints), swollen joints (28 joints), patient's global assessment of disease activity, physician's global assessments of disease activity, and CRP. The total score range is from 0 to 86 with a lower score indicating less disease activity. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Units on a Scale
  Change at Week 2 | -4.5129 (9.68032) | -9.1095 (9.64598) | -7.9649 (9.58765)
  Change at Week 4 | -7.3134 (11.87959) | -13.3976 (12.00410) | -12.2156 (11.65262)
  Change at Week 6 | -9.5833 (13.15531) | -16.1013 (12.80166) | -15.4404 (12.18642)
  Change at Week 8 | -10.0752 (13.54599) | -17.6624 (12.98109) | -17.1302 (12.92830)
  Change at Week 12 | -11.5975 (14.53181) | -19.6639 (13.67016) | -19.0635 (13.63444)
  Change at Week 16 | -11.3507 (15.72864) | -20.3221 (14.14177) | -20.0652 (13.85171)
  Change at Week 18 | -10.6805 (16.31549) | -20.1215 (14.75683) | -20.4858 (13.72370)
  Change at Week 20 | -11.0425 (16.42770) | -20.8300 (15.31245) | -20.8508 (14.44400)
  Change at Week 24 | -11.1443 (16.37909) | -20.7459 (15.48312) | -21.0858 (14.57962)
  Change at Week 28 | -11.7828 (17.04652) | -21.3535 (15.98762) | -21.5524 (14.69362)
  Change at Week 32 | -12.0835 (17.11297) | -21.8176 (16.15549) | -21.8530 (14.58393)
  Change at Week 36 | -12.2107 (17.24703) | -21.9077 (15.95251) | -22.1040 (14.54871)
  Change at Week 40 | -11.9185 (17.32206) | -21.7862 (16.12260) | -21.6692 (15.33635)
  Change at Week 44 | -11.8730 (17.41934) | -21.4843 (16.33985) | -21.5514 (15.78476)
  Change at Week 48 | -11.9055 (17.91398) | -21.7238 (16.45520) | -21.7991 (15.34514)
  Change at Week 52 | -11.7647 (17.61074) | -21.9130 (16.32611) | -21.7344 (15.64620)

15. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score Through Week 52
Description: The CDAI score is a derived score of 4 components: tender joints (28 joints), swollen joints (28 joints), patient's global assessment of disease activity, and physician's global assessments of disease activity. The total score ranges from 0 to 76 with a lower score indicating less disease activity. A negative change in CDAI score indicates an improvement in disease activity and a positive change in score indicates a worsening of disease activity. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Units on a Scale
  Change at Week 2 | -4.38 (9.210) | -6.82 (9.350) | -5.65 (9.014)
  Change at Week 4 | -7.09 (11.241) | -11.13 (11.699) | -9.88 (11.166)
  Change at Week 6 | -9.24 (12.407) | -13.79 (12.416) | -13.10 (11.599)
  Change at Week 8 | -9.72 (12.714) | -15.37 (12.593) | -14.79 (12.438)
  Change at Week 12 | -11.19 (13.625) | -17.36 (13.223) | -16.74 (13.098)
  Change at Week 16 | -10.86 (14.716) | -18.04 (13.651) | -17.75 (13.261)
  Change at Week 18 | -10.24 (15.245) | -17.82 (14.291) | -18.17 (13.204)
  Change at Week 20 | -10.57 (15.338) | -18.53 (14.809) | -18.57 (13.910)
  Change at Week 24 | -10.68 (15.302) | -18.45 (14.936) | -18.80 (14.075)
  Change at Week 28 | -11.27 (15.926) | -19.06 (15.395) | -19.27 (14.168)
  Change at Week 32 | -11.55 (15.950) | -19.57 (15.549) | -19.56 (14.095)
  Change at Week 36 | -11.70 (16.099) | -19.66 (15.455) | -19.80 (14.084)
  Change at Week 40 | -11.46 (16.236) | -19.54 (15.640) | 19.3 (14.833)
  Change at Week 44 | -11.41 (16.126) | -19.24 (15.888) | -19.26 (15.264)
  Change at Week 48 | -11.47 (16.594) | -19.47 (15.951) | -19.50 (14.871)
  Change at Week 52 | -11.38 (16.348) | -19.67 (15.834) | -19.44 (15.115)

16. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index Based (SDAI-based) American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) Remission Through Week 52
Description: Participant having SDAI-based ACR/EULAR remission at a visit if SDAI score is of <= 3.3. SDAI derived by combining 5 disease assessments: tender joint (28), swollen joint (28) counts, participants global assessment of disease activity using VAS (scale ranges from 0 to 10 [0 =very well to 10 = very poor]), physicians global assessment of disease activity using VAS (scale ranges from 0 to 10 [0=no arthritis to 10=extremely active arthritis]) and CRP. 28 joints evaluated for swelling and tenderness are same set of 28 joints used in DAS28 includes shoulder, elbow, wrist, MCP1, MCP2, MCP3, MCP4, MCP5, PIP1, PIP2, PIP3, PIP4, PIP5 joints of upper right and left extremities and knee joints of lower right and left extremities. Change from baseline in SDAI score measures change in disease activity, where negative change= improvement and positive change= worsening. Participants were analyzed according to randomized treatment groups they were assigned regardless of treatments actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: Full analysis set included all randomized participants. Participants were set to not achieving SDAI-based remission after meeting EE, LE or TF criteria (whichever is earliest) or if having data missing.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 0.2 | 0 | 0
  Week 4 | 0.4 | 0.2 | 1.3
  Week 6 | 0.4 | 1.6 | 2.3
  Week 8 | 0.7 | 2.9 | 2.9
  Week 12 | 1.6 | 4.8 | 5.2
  Week 16 | 2.2 | 5.4 | 6.6
  Week 18 | 1.6 | 6.3 | 6.8
  Week 20 | 1.6 | 7.5 | 7.7
  Week 24 | 2.3 | 8.1 | 9.5
  Week 28 | 2.3 | 9.0 | 8.4
  Week 32 | 2.9 | 9.7 | 10.2
  Week 36 | 1.8 | 10.1 | 10.6
  Week 40 | 2.5 | 11.5 | 11.5
  Week 44 | 2.5 | 9.7 | 11.7
  Week 48 | 3.8 | 11.3 | 10.4
  Week 52 | 3.2 | 11.5 | 10.6

17. Secondary Outcome: Percentage of Participants With Boolean-based American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) Remission Through Week 52
Description: A participant was considered as having achieved the Boolean-based American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) remission at a visit if all of the following 4 criteria were met at that visit: Tender joint count (68 joints) less than or equal to (<=) 1; Swollen joint count (66 joints) <=1; CRP <=1 milligram per deciliter (mg/dL); Patient's Global Assessment of Disease Activity <=1 on a 0 (very well) to 10 (very poor) VAS. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: Full analysis set included all randomized participants. Participants were set to not achieving Boolean-based remission after meeting EE, LE or TF criteria (whichever is earliest) or if having data missing.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 0.2 | 0.4 | 0
  Week 4 | 0.2 | 0.4 | 0.7
  Week 6 | 0 | 0.9 | 0.9
  Week 8 | 0.2 | 1.3 | 1.8
  Week 12 | 1.3 | 2.9 | 3.1
  Week 16 | 1.6 | 3.2 | 4.7
  Week 18 | 0.7 | 3.6 | 4.7
  Week 20 | 1.3 | 4.3 | 5.6
  Week 24 | 0.9 | 4.3 | 7.0
  Week 28 | 1.1 | 5.2 | 6.1
  Week 32 | 2.3 | 5.0 | 6.5
  Week 36 | 1.3 | 7.0 | 7.9
  Week 40 | 0.9 | 5.9 | 7.9
  Week 44 | 1.4 | 5.7 | 7.9
  Week 48 | 1.8 | 7.0 | 7.0
  Week 52 | 2.2 | 7.0 | 5.7

18. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score Through Week 52
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) score is an evaluation of the functional status for a participant. The 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Negative change reflects an improvement and a positive change reflects a worsening. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 18, 20, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Units on a Scale
  Change at Week 2 | -0.075 (0.3809) | -0.139 (0.3744) | -0.128 (0.3939)
  Change at Week 4 | -0.130 (0.4444) | -0.244 (0.4498) | -0.254 (0.4184)
  Change at Week 6 | -0.170 (0.4657) | -0.318 (0.4989) | -0.360 (0.4910)
  Change at Week 8 | -0.172 (0.4824) | -0.362 (0.5163) | -0.388 (0.5163)
  Change at Week 12 | -0.191 (0.5055) | -0.387 (0.5512) | -0.399 (0.5364)
  Change at Week 16 | -0.201 (0.5439) | -0.409 (0.5736) | -0.433 (0.5489)
  Change at Week 18 | -0.217 (0.5266) | -0.431 (0.5744) | -0.464 (0.5496)
  Change at Week 20 | -0.209 (0.5275) | -0.429 (0.6074) | -0.474 (0.5797)
  Change at Week 28 | -0.232 (0.5515) | -0.438 (0.5837) | -0.471 (0.5763)
  Change at Week 32 | -0.225 (0.5462) | -0.441 (0.6017) | -0.483 (0.5886)
  Change at Week 36 | -0.226 (0.5585) | -0.444 (0.5961) | -0.461 (0.5810)
  Change at Week 40 | -0.230 (0.5586) | -0.447 (0.5900) | -0.431 (0.5921)
  Change at Week 44 | -0.228 (0.5601) | -0.442 (0.6182) | -0.456 (0.5956)
  Change at Week 48 | -0.227 (0.5727) | -0.447 (0.6207) | -0.481 (0.6043)
  Change at Week 52 | -0.225 (0.5693) | -0.453 (0.6127) | -0.470 (0.5959)

19. Secondary Outcome: Area Under the Curve (AUC) of Change From Baseline in HAQ-DI Score From Week 0 Through Week 24 and From Week 0 Through Week 52
Description: HAQ-DI has 20-question in 8 functional areas: dressing, arising, eating, walking, hygiene, reaching, gripping, and daily living activities, scored from 0=no difficulty to 3=inability to perform task in that area. Overall score computed as sum of domain score divided by number of domains answered. Total possible score range 0= least difficulty to 3= extreme difficulty. AUC of change from baseline in HAQ-DI score is AUC of change from baseline in HAQ-DI score versus time. AUC was calculated based on measurement (observed HAQ-DI score change from baseline) at scheduled visits using trapezoidal rule.Functional status was determined as cumulative measure of HAQ-DI over 1 year by using AUC of change from baseline in HAQ-DI score through week 52. Decreases in AUC of change from baseline in HAQ-DI means greater average improvement in physical function over time. Participants analyzed according to randomized treatment groups they were assigned, regardless of treatments they actually received.
Time Frame: Week 0 Through Week 24 and 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a Scale*Day
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Units on a Scale*Day
  Week 0 Through Week 24 | -28.85 (69.783) | -57.99 (76.384) | -61.71 (75.189)
  Week 0 Through Week 52 | -73.55 (170.636) | -145.30 (184.630) | -153.03 (180.633)

20. Secondary Outcome: Percentage of Participants With Health Assessment Questionnaire-Disability Index (HAQ-DI) Response Through Week 52
Description: HAQ-DI response was defined as change of less than -0.22 from baseline in HAQ-DI score. The HAQ-DI score is an evaluation of the functional status for a participant. The 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 34.4 | 40.6 | 37.0
  Week 4 | 38.1 | 49.2 | 52.2
  Week 6 | 42.4 | 56.2 | 58.0
  Week 8 | 44.1 | 56.2 | 61.0
  Week 12 | 44.6 | 60.1 | 60.9
  Week 16 | 45.5 | 60.9 | 61.9
  Week 18 | 45.9 | 62.7 | 65.4
  Week 20 | 46.2 | 61.4 | 65.4
  Week 24 | 46.9 | 63.0 | 65.4
  Week 28 | 47.8 | 64.8 | 63.4
  Week 32 | 46.9 | 62.8 | 63.7
  Week 36 | 47.3 | 63.9 | 63.7
  Week 40 | 47.3 | 63.7 | 61.8
  Week 44 | 47.3 | 62.1 | 63.2
  Week 48 | 47.3 | 61.8 | 64.6
  Week 52 | 47.1 | 63.4 | 64.5

21. Secondary Outcome: Percentage of Participants With Health Assessment Questionnaire-Disability Index (HAQ-DI) Score of Less Than or Equal to 0.5
Description: HAQ-DI score is an evaluation of the functional status for a participant. The 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 2 | 7.9 | 12.2 | 11.5
  Week 4 | 9.9 | 15.6 | 16.3
  Week 6 | 9.5 | 18.3 | 21.2
  Week 8 | 10.6 | 21.7 | 21.0
  Week 12 | 12.2 | 22.8 | 23.3
  Week 16 | 13.3 | 24.6 | 26.8
  Week 18 | 13.7 | 24.6 | 25.9
  Week 20 | 13.1 | 26.0 | 27.5
  Week 24 | 13.1 | 25.9 | 27.5
  Week 28 | 13.8 | 26.2 | 28.7
  Week 32 | 13.7 | 26.0 | 28.7
  Week 36 | 13.7 | 27.5 | 27.5
  Week 40 | 13.7 | 27.3 | 26.2
  Week 44 | 13.1 | 27.8 | 27.6
  Week 48 | 13.8 | 28.2 | 30.0
  Week 52 | 12.4 | 27.5 | 29.3

22. Secondary Outcome: Change From Baseline in Van Der Heijde-modified Sharpe (vdH-S) Score at Week 24
Description: vdH-S score is defined as a measurement of progression in structural damage. It is the sum of joint erosion (32 joints of the hands and 12 joints of the feet) score and joint space narrowing (JSN) (30 joints of the hands and 12 joints of the feet) score. The joint erosion assessment is scored according to the surface area involved, from 0 to 5, with 0 indicating no erosion and 5 indicating complete collapse of bone whereas the JSN assessment including subluxation, is scored from 0 (normal) to 4 (bony ankylosis or complete luxation). The total score ranges from 0 (best) to 448 (worst) with higher scores indicating more joint damage. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 550 | 553 | 551
Units on a Scale | 1.96 (5.390) | 0.35 (2.149) | 0.30 (2.165)

23. Secondary Outcome: Change From Baseline in Van Der Heijde-modified Sharpe (vdH-S) Sub-score by Type of Damage (Erosion or JSN) at Week 24 and 52
Description: vdH-S score measures structural damage progression as sum of joint erosion(JE) and joint space narrowing(JSN) scores(S).JE is summary of erosion severity in 32 of hands(H) and 12 of feet(F) joints, scored as per surface area- from 0 (no erosion) to 5 (complete(CM) collapse of bone). Maximum (MAX) JES for H-160 (32*5) and MAX JES for F- 120 (12*10 [5*2 sides of foot]). MAX JES is 280 whereas JSN is summary of severity of 30 of H and 12 of F joints, scored to subluxation from 0(normal) to 4(bony ankylosis or CM luxation). MAX JSNS for H-120(30*4), and MAX JSS for F-48(12*4). MAX JSNS is 168.Thus MAX JES-280 combined with MAX JSNS-168 gives worst possible vdH-SS (i.e., JE score + JSN score) of 448. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 550 | 553 | 551
Units on a Scale
  Erosion Score: Change at Week 24 | 1.21 (3.348) | 0.10 (1.306) | 0.08 (1.321)
  JSN Score: Change at Week 24 | 0.76 (2.540) | 0.24 (1.404) | 0.21 (1.537)
  Erosion Score: Change at Week 52 | 2.23 (5.903) | 0.12 (1.809) | 0.08 (2.005)
  JSN Score: Change at Week 52 | 1.46 (4.311) | 0.38 (1.839) | 0.38 (2.184)

24. Secondary Outcome: Change From Baseline in Van Der Heijde-modified Sharpe (vdH-S) Sub-score by Region Hand or Feet and Type Erosion or JSN at Week 24 and 52
Description: vdH-S score measures structural damage progression as sum of joint erosion(JE) and joint space narrowing(JSN) scores(S).JE is summary of erosion severity in 32 of hands(H) and 12 of feet(F) joints, scored as per surface area- from 0 (no erosion) to 5 (complete(CM) collapse of bone). Maximum (MAX) JES for H-160 (32*5) and MAX JES for F- 120 (12*10 [5*2 sides of foot]). MAX JES is 280 whereas JSN is summary of severity of 30 of H and 12 of F joints, scored to subluxation from 0(normal) to 4(bony ankylosis or CM luxation). MAX JSNS for H-120(30*4), and MAX JSS for F-48(12*4). MAX JSNS is 168.Thus MAX JES-280 combined with MAX JSNS-168 gives worst possible vdH-SS (i.e., erosion score + JSN score) of 448. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 550 | 553 | 551
Units on a Scale
  Change in Hand Erosion Score at Week 24 | 0.74 (2.406) | 0.07 (0.920) | 0.03 (0.966)
  Change in Hand JSN Score at Week 24 | 0.51 (1.818) | 0.16 (1.025) | 0.16 (1.021)
  Change in Foot Erosion Score at Week 24 | 0.46 (1.459) | 0.03 (0.682) | 0.05 (0.754)
  Change in Foot JSN Score at Week 24 | 0.25 (1.207) | 0.09 (0.722) | 0.06 (1.152)
  Change in Hand Erosion Score at Week 52 | 1.43 (4.378) | 0.09 (1.296) | 0.03 (1.312)
  Change in Hand JSN Score at Week 52 | 0.98 (3.196) | 0.25 (1.378) | 0.28 (1.808)
  Change in Foot Erosion Score at Week 52 | 0.80 (2.460) | 0.03 (0.955) | 0.06 (1.302)
  Change in Foot JSN Score at Week 52 | 0.48 (2.013) | 0.13 (0.929) | 0.10 (1.171)

25. Secondary Outcome: Percentage of Participants With Change From Baseline in Van Der Heijde Modified Sharpe Score (vdH-S Score) Greater Than Smallest Detectable Change (SDC) at Weeks 24 and 52
Description: vdH-S score measures structural damage progression as sum of joint erosion(JE) and joint space narrowing(JSN) scores(S). JE is summary of erosion severity in 32 of hand and 12 of feet joints, scored according to the surface area, from 0 (no erosion) to 5 (complete collapse of bone) whereas the JSN is summary of severity of 30 of hand and 12 of feet joints, scored according to the subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation). The SDC is smallest change in score that is considered to be assessed correctly based on limits of agreement (that is., above the measurement error). The SDC for change from baseline in vdH-S Score is determined as: SDC=1.96 * SD / (root 2 * root k), where SD is the standard deviation of the difference between 2 readers in change from baseline in vdH-S score; k is the number of readers. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Weeks 24 and 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 550 | 553 | 551
Percentage of Participants
  Week 24 | 25.3 | 8.3 | 7.6
  Week 52 | 35.5 | 12.1 | 12.0

26. Secondary Outcome: Percentage of Participants With a Change of Less Than or Equal to 0 From Baseline in Van Der Heijde Modified Sharpe (vdH-S) Score at Weeks 24 and 52
Description: vdH-S score measures structural damage progression as sum of joint erosion(JE) and joint space narrowing(JSN) scores(S).JE is summary of erosion severity in 32 of hands(H) and 12 of feet(F) joints, scored as per surface area- from 0 (no erosion) to 5 (complete(CM) collapse of bone). Maximum (MAX) JES for H-160 (32*5) and MAX JES for F- 120 (12*10 [5*2 sides of foot]). MAX JES is 280 whereas JSN is summary of severity of 30 of H and 12 of F joints, scored to subluxation from 0(normal) to 4(bony ankylosis or CM luxation). MAX JSNS for H-120(30*4), and MAX JSS for F-48(12*4). MAX JSNS is 168.Thus MAX JES-280 combined with MAX JSNS-168 gives worst possible vdH-SS of (i.e., erosion score + JSN score) 448. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 24 and 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 550 | 553 | 551
Percentage of Participants
  Week 24 | 48.4 | 65.8 | 68.8
  Week 52 | 45.5 | 59.0 | 62.4

27. Secondary Outcome: Change From Baseline in Van Der Heijde Modified Sharpe Score (vdH-S Score) by Reader at Weeks 24 and 52
Description: as for outcome 23
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 550 | 553 | 551
Units on a Scale
  Reader 1 at Week 24: number analyzed (Participants) | 550 | 551 | 550
  Reader 1 at Week 24 | 2.06 (5.616) | 0.21 (2.495) | 0.20 (2.773)
  Reader 2 at Week 24 | 1.65 (5.053) | 0.38 (1.969) | 0.33 (1.830)
  Reader 1 at Week 52: number analyzed (Participants) | 447 | 459 | 467
  Reader 1 at Week 52 | 2.99 (7.940) | 0.54 (3.285) | 0.29 (3.325)
  Reader 2 at Week 52: number analyzed (Participants) | 447 | 460 | 467
  Reader 2 at Week 52 | 2.65 (7.331) | 0.54 (2.660) | 0.35 (2.184)

28. Secondary Outcome: Change From Baseline in Serum C-reactive Protein (CRP) Levels Through Week 52
Description: Serum CRP is a marker of systemic inflammation. A negative change from baseline in CRP represents improvement. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: Full analysis set included all randomized participants. Last Observation Carried Forward (LOCF) method was used to impute missing values. The last observation at or prior to EE/LE was used to replace the data after EE/LE for participants who met EE/LE criteria.
Measure: Mean (Standard Deviation); unit: Milligram per Deciliter
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Milligram per Deciliter
  Baseline | 2.5148 (3.38577) | 2.4145 (2.62179) | 2.3952 (2.64241)
  Change at Week 2 | -0.1339 (2.86946) | -2.2867 (2.44604) | -2.3198 (2.64772)
  Change at Week 4 | -0.2209 (2.94279) | -2.2707 (2.41525) | -2.3406 (2.64584)
  Change at Week 6 | -0.3432 (2.96865) | -2.3124 (2.44604) | -2.3451 (2.64678)
  Change at Week 8 | -0.3561 (3.05281) | -2.2919 (2.41368) | -2.3392 (2.65864)
  Change at Week 12 | -0.4099 (3.22085) | -2.3038 (2.43828) | -2.3274 (2.67383)
  Change at Week 16 | -0.4890 (3.17554) | -2.2841 (2.43707) | -2.3166 (2.65115)
  Change at Week 18 | -0.4375 (3.48359) | -2.3030 (2.45255) | -2.3114 (2.65919)
  Change at Week 20 | -0.4682 (3.21483) | -2.2973 (2.44855) | -2.2798 (2.74939)
  Change at Week 24 | -0.4610 (3.31445) | -2.2974 (2.45343) | -2.2891 (2.73480)
  Change at Week 28 | -0.5108 (3.34288) | -2.2937 (2.45419) | -2.2820 (2.73435)
  Change at Week 32 | -0.5332 (3.39542) | -2.2474 (2.63824) | -2.2907 (2.73375)
  Change at Week 36 | -0.5128 (3.36374) | -2.2515 (2.62647) | -2.3085 (2.73396)
  Change at Week 40 | -0.4623 (3.46179) | -2.2429 (2.64450) | -2.3032 (2.73402)
  Change at Week 44 | -0.4631 (4.00446) | -2.2398 (2.65898) | -2.2895 (2.75035)
  Change at Week 48 | -0.4372 (4.15311) | -2.2561 (2.62491) | -2.2944 (2.75776)
  Change at Week 52 | -0.3854 (3.96633) | -2.2399 (2.64267) | -2.2976 (2.73878)

29. Secondary Outcome: Change From Baseline in the Duration of Morning Stiffness Through Week 52
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (If none was present = 0; If morning stiffness was continuing at the time of assessment or was unusual compared to the recent past, average of duration of stiffness over the past 3 days was reported; If stiffness persisted the entire day, 1440 minutes was recorded). Negative values for this outcome measure represent improvement, i.e. shortening of duration of morning stiffness. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: Full analysis set was defined as all randomized participants. Here 'N'(number of participants analyzed): Evaluable for this outcome measure. Last Observation Carried Forward (LOCF) method was used to impute missing values. The last observation at or prior to EE/LE was used to replace the data after EE/LE for participants who met EE/LE criteria.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 552 | 552 | 555
Minutes
  Change at Week 2 | -22.5 (184.96) | -35.2 (212.94) | -24.0 (177.41)
  Change at Week 4 | -27.2 (202.02) | -61.6 (213.09) | -45.1 (181.13)
  Change at Week 6 | -35.3 (190.54) | -81.0 (207.07) | -70.3 (206.41)
  Change at Week 8 | -41.7 (171.05) | -84.1 (232.34) | -79.6 (213.42)
  Change at Week 12 | -53.2 (179.24) | -88.1 (220.03) | -89.4 (217.48)
  Change at Week 16 | -52.2 (173.24) | -82.2 (241.75) | -84.1 (224.72)
  Change at Week 18 | -60.2 (191.68) | -84.6 (239.43) | -88.5 (223.95)
  Change at Week 20 | -62.0 (193.64) | -93.5 (234.10) | -90.0 (229.08)
  Change at Week 24 | -63.7 (195.58) | -96.7 (228.31) | -95.5 (234.19)
  Change at Week 28 | -68.3 (195.42) | -95.2 (230.36) | -98.0 (235.03)
  Change at Week 32 | -68.9 (196.31) | -96.5 (230.46) | -96.5 (231.25)
  Change at Week 36 | -68.8 (196.90) | -96.5 (228.71) | -95.2 (226.37)
  Change at Week 40 | -68.7 (197.06) | -95.7 (243.78) | -95.9 (233.28)
  Change at Week 44 | -69.9 (197.38) | -96.6 (232.42) | -97.0 (234.63)
  Change at Week 48 | -69.6 (195.50) | -97.8 (238.36) | -97.0 (230.66)
  Change at Week 52 | -67.3 (196.98) | -99.1 (233.82) | -97.7 (231.53)

30. Secondary Outcome: Change From Baseline in Physical and Mental Component Summary Scores of 36-Item Short Form Health Survey (SF-36) at Weeks 24 and 52
Description: SF-36 questionnaire is health related quality of life (QOL) instrument with 36 questions with 8 multi-item scales (evaluated limitations in): physical functioning due to health problems; usual role activities due to physical health problems; Bodily pain; General mental health (psychological distress and well-being); usual role activities due to personal or emotional problems; social functioning due to physical or mental health problems; Vitality (energy and fatigue); General health perception. Each 8 scales scored from 0 to 100 with higher scores= better health. Based on scale scores, summary scores, physical component score (PCS) and mental component score (MCS) will be derived. Scoring is derived based on algorithm developed in software provided by developer. Summary MCS and PCS score is also scaled from 0 to 100 with higher scores= better health. Participants were analyzed according to randomized treatment groups they were assigned regardless of treatments they actually received.
Time Frame: Baseline, Week 24 and 52
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Units on a Scale
  PCS :Change at Week 24 | 2.290 (6.2790) | 5.358 (7.3312) | 5.850 (7.0677)
  PCS :Change at Week 52 | 2.423 (6.8069) | 5.661 (7.7405) | 6.162 (7.2277)
  MCS :Change at Week 24 | 2.892 (9.1766) | 4.898 (9.6508) | 4.216 (9.4819)
  MCS :Change at Week 52 | 2.690 (9.5698) | 5.351 (9.6397) | 4.767 (9.7991)

31. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 4-Point Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 8, 16, 24, 36 and 52
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The questionnaire consists of 13 questions that assess a participant's level of fatigue and tiredness over the last 7 days. Each question is graded on a 5-point scale (0 - 4); and accordingly, the total FACIT-Fatigue scores can range from 0 to 52, with lower score reflecting more fatigue and higher scores reflecting less fatigue. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Week 8, 16, 24, 36 and 52
Population: as for outcome 28
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Percentage of Participants
  Week 8 | 41.0 | 55.8 | 54.9
  Week 16 | 42.4 | 58.0 | 58.9
  Week 24 | 43.9 | 61.4 | 59.4
  Week 36 | 39.7 | 57.8 | 56.2
  Week 52 | 41.0 | 59.1 | 60.5

32. Secondary Outcome: Change From Baseline in Total Scores of Work Limitations Questionnaire (WLQ) Week 8, 16, 24, 36 and 52
Description: The Work Limitations Questionnaire (WLQ) was used to measure the impairment in work-related productivity, with reference to the previous two weeks. Each work-related question is scored from 0 to 4 and the total score ranges from 0-100, with lower scores signifying fewer limitations at work. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 8, 16, 24, 36 and 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 227 | 223 | 223
Units on a Scale
  Week 8 | -0.812 (3.6230) | -1.946 (3.8040) | -2.202 (3.8437)
  Week 16 | -0.840 (4.6414) | -2.406 (4.1403) | -2.600 (4.3066)
  Week 24 | -1.019 (4.5328) | -2.765 (4.4381) | -2.884 (4.5873)
  Week 36 | -0.940 (4.7982) | -2.921 (4.4205) | -2.952 (4.5640)
  Week 52 | -0.732 (5.0288) | -3.057 (4.5290) | -2.936 (4.3940)

33. Secondary Outcome: Change From Baseline in EuroQol Health State Visual Analogue Scale (EQ VAS)
Description: The EuroQol Health State Visual Analogue Scale (EQ VAS) records the respondent's self-rated health on a vertical line, VAS where the endpoints are labeled as 0= 'Worst imaginable health state' and 100= 'Best imaginable health state'. The EQ VAS can be used as a quantitative measure of health outcome as judged by the individual respondents. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: Baseline, Week 8, 16, 24, 36 and 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 554 | 557 | 556
Units on a Scale
  Change at Week 8 | 5.61 (24.415) | 11.64 (26.979) | 12.24 (26.025)
  Change at Week 16 | 5.83 (26.177) | 14.09 (28.581) | 14.36 (27.884)
  Change at Week 24 | 6.71 (26.520) | 14.86 (28.747) | 16.41 (28.830)
  Change at Week 52 | 8.30 (26.144) | 16.80 (28.595) | 17.14 (28.329)

34. Secondary Outcome: Change From Baseline in EuroQol EQ-5D-3L Descriptive System
Description: The EQ-5D-3L Descriptive System comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead. Participants were analyzed according to the randomized treatment groups they were assigned to, regardless of the treatments they actually received.
Time Frame: at Week 8, 16, 24, and 52
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 556 | 557 | 557
Units on a Scale
  Change at Week 8 | 0.1041 (0.31794) | 0.1734 (0.32473) | 0.1647 (0.30146)
  Change at Week 16 | 0.1131 (0.33788) | 0.1831 (0.34875) | 0.1899 (0.31149)
  Change at Week 24 | 0.1263 (0.33539) | 0.1885 (0.33867) | 0.2057 (0.32081)
  Change at Week 52 | 0.1255 (0.34312) | 0.1950 (0.33448) | 0.2007 (0.32895)

ADVERSE EVENTS:
Time Frame: Screening up to Week 120
Description: Safety population included all participants received at least 1 partial or complete dose of study drug and analyzed in the treatment they actually received over study period, regardless of the treatments they were randomized to. One Participant randomized to sirukumab 50 mg but inadvertently received 1 dose of 100 mg at week 16. The participant was included in 100 mg group for safety, due to which total participants increased by 1 in 100 mg group (558) and decreased by 1 in 50 mg group (556).
Groups:
- Week 0 to Week 120-Placebo: Participants received matching placebo from week 0 to week 50, every 2 weeks (q2w) until either early escape (EE) at Week 18 or late escape (LE) at Week 40 or crossover (CO) at Week 52 and were rerandomized to subcutaneous (SC) sirukumab 50 mg q4w or sirukumab 100 mg q2w dose regimens up to Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
- W0 to W120-Placebo to Sirukumab 50 mg q4w Due to EE/LE or CO: Participants who received placebo in the placebo controlled period were rerandomized (due to EE at Week 18 or LE at Week 40 or CO at Week 52) to receive subcutaneous (SC) sirukumab 50 mg q4w dose regimen up to Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
- W0 to W120- Sirukumab 50 mg q4w: Participants received 50 mg of sirukumab SC injections at Weeks 0, 4, and q4w through Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
- W0 to W120- Placebo to Sirukumab 100 mg q2w Due to EE/LE or CO: Participants who received placebo in the placebo controlled period were rerandomized (due to EE at Week 18 or LE at Week 40 or CO at Week 52) to receive subcutaneous (SC) sirukumab 100 mg q2w dose up to Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
- W0 to W120-Sirukumab 100 mg q2w: Participants received 100 mg of sirukumab SC injections at Weeks 0, 2 and q2w throught Week 104. Participants who completed study agent administration up to Week 104 and did not elect for long term extension (LTE) were followed up for safety from Week 104 up to Week 120.
Arm/Group | Week 0 to Week 120-Placebo | W0 to W120-Placebo to Sirukumab 50 mg q4w Due to EE/LE or CO | W0 to W120- Sirukumab 50 mg q4w | W0 to W120- Placebo to Sirukumab 100 mg q2w Due to EE/LE or CO | W0 to W120-Sirukumab 100 mg q2w
Serious Adverse Events (participants affected / at risk) | 40/556 | 30/242 | 111/556 | 35/241 | 97/558
Other Adverse Events (participants affected / at risk) | 213/556 | 113/242 | 355/556 | 128/241 | 353/558
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Week 0 to Week 120-Placebo (N=556) | W0 to W120-Placebo to Sirukumab 50 mg q4w Due to EE/LE or CO (N=242) | W0 to W120- Sirukumab 50 mg q4w (N=556) | W0 to W120- Placebo to Sirukumab 100 mg q2w Due to EE/LE or CO (N=241) | W0 to W120-Sirukumab 100 mg q2w (N=558)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Acute Left Ventricular Failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 3 | 1 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Basedow's Disease (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Amaurosis Fugax (Eye disorders) | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Scleritis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 2 | 0 | 0
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diverticular Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Enterocele (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Erosive Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric Polyps (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis Erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatic Fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 1 | 1 | 0 | 2
Death (General disorders) | 0 | 0 | 1 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 1
Medical Device Site Joint Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Serositis (General disorders) | 0 | 1 | 0 | 0 | 0
Sudden Cardiac Death (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 3
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 3
Gallbladder Perforation (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic Cyst (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Non-Alcoholic Steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abdominal Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 3 | 0 | 4
Abscess Soft Tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Appendicitis Perforated (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bacterial Food Poisoning (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 7 | 2 | 5
Cellulitis Staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cytomegalovirus Colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Dengue Fever (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Device Related Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 4 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Escherichia Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Extradural Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Eye Infection Fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hepatitis E (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infected Bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infectious Pleural Effusion (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Infective Spondylitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Intervertebral Discitis (Infections and infestations) | 0 | 1 | 1 | 1 | 1
Localised Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 2 | 0 | 2
Osteomyelitis Chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Perirectal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 2 | 3 | 0 | 0
Peritonsillar Abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 11 | 1 | 10
Pneumonia Bacterial (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Pneumonia Necrotising (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Post Procedural Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyonephrosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Salpingo-Oophoritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 3 | 1 | 5
Septic Shock (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1 | 1 | 3
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abdominal Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Chemical Peritonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Epiphyseal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Joint Capsule Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Kidney Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 5
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 1 | 3
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 2 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 2 | 0
Chest X-Ray Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Liver Function Test Increased (Investigations) | 1 | 0 | 0 | 1 | 1
Weight Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Atlantoaxial Instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Fistula Discharge (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 1 | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 0 | 5 | 1 | 5
Rheumatoid Nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Benign Neoplasm of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Intraductal Papilloma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Neuroendocrine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Oropharyngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ovarian Clear Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Cervical Myelopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cervical Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Hypertensive Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Intracranial Aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Pyramidal Tract Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Reversible Cerebral Vasoconstriction Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Trigeminal Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ulnar Nerve Palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Blighted Ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Device Dislocation (Product Issues) | 0 | 0 | 0 | 0 | 1
Device Failure (Product Issues) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 3 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1 | 1 | 0
Breast Mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary Necrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Aortic Dissection (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Axillary Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Extremity Necrosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Labile Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Necrosis Ischaemic (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Thrombosed Varicose Vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Week 0 to Week 120-Placebo (N=556) | W0 to W120-Placebo to Sirukumab 50 mg q4w Due to EE/LE or CO (N=242) | W0 to W120- Sirukumab 50 mg q4w (N=556) | W0 to W120- Placebo to Sirukumab 100 mg q2w Due to EE/LE or CO (N=241) | W0 to W120-Sirukumab 100 mg q2w (N=558)
Leukopenia (Blood and lymphatic system disorders) | 7 | 12 | 37 | 8 | 39
Neutropenia (Blood and lymphatic system disorders) | 5 | 9 | 40 | 8 | 34
Diarrhoea (Gastrointestinal disorders) | 21 | 2 | 28 | 9 | 23
Injection Site Erythema (General disorders) | 6 | 11 | 50 | 31 | 70
Injection Site Pruritus (General disorders) | 1 | 3 | 12 | 14 | 34
Injection Site Swelling (General disorders) | 0 | 3 | 15 | 13 | 27
Bronchitis (Infections and infestations) | 27 | 17 | 48 | 13 | 36
Nasopharyngitis (Infections and infestations) | 53 | 16 | 70 | 19 | 67
Pharyngitis (Infections and infestations) | 13 | 5 | 30 | 8 | 24
Upper Respiratory Tract Infection (Infections and infestations) | 63 | 28 | 76 | 20 | 72
Urinary Tract Infection (Infections and infestations) | 13 | 8 | 30 | 13 | 23
Alanine Aminotransferase Increased (Investigations) | 23 | 34 | 108 | 41 | 124
Aspartate Aminotransferase Increased (Investigations) | 17 | 20 | 63 | 23 | 84
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 36 | 9 | 46 | 10 | 29
Headache (Nervous system disorders) | 22 | 8 | 38 | 9 | 28
Hypertension (Vascular disorders) | 21 | 14 | 32 | 11 | 45

LIMITATIONS AND CAVEATS:
The short pure placebo-controlled period (through Week 18) and the EE at Week 18 and LE at Week 40 for participants in the placebo group might have affected the ability to directly compare safety between sirukumab and placebo groups through Week 52.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.